CLINICAL TRIAL: NCT05134974
Title: Randomized, Parallel Arm, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) to Reverse Pharmacologically-Induced Mydriasis in Healthy Subjects
Brief Title: Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) to Reverse Pharmacologically-Induced Mydriasis (MIRA-3)
Acronym: MIRA-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPI-NYXRM-302 (MIRA-3)
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Mydriasis; Dilation
Keywords: Nyxol; Pharmacologically Induced Mydriasis; Dilation
MeSH Terms: conditions — Mydriasis; Dilatation, Pathologic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentolamine Ophthalmic Solution 0.75% (Active Comparator): 2 drops in study eye and 1 drop in non-study eye, 1 hour post pharmacologically-induced mydriasis
  Interventions: Drug: Phentolamine Ophthalmic Solution 0.75%
- Phentolamine Ophthalmic Solution Vehicle (Placebo Comparator): 2 drops in study eye and 1 drop in non-study eye, 1 hour post pharmacologically-induced mydriasis
  Interventions: Drug: Phentolamine Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: Phentolamine Ophthalmic Solution 0.75% — 0.75% phentolamine ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol®; Nyxol
  Arms: Phentolamine Ophthalmic Solution 0.75%
Drug: Phentolamine Ophthalmic Solution Vehicle — Phentolamine Ophthalmic Solution Vehicle
  Arms: Phentolamine Ophthalmic Solution Vehicle

SUMMARY:
The objectives of this study are:

* To evaluate the efficacy of Nyxol to expedite the reversal of pharmacologically-induced mydriasis across multiple mydriatic agents with an emphasis on phenylephrine
* To evaluate the efficacy of Nyxol to return subjects to baseline accommodation after worsening (with cycloplegic agents tropicamide and Paremyd)
* To evaluate the safety of Nyxol
* To evaluate any additional benefits of the reversal of pharmacologically-induced mydriasis
* To evaluate the systemic exposure of Nyxol on pharmacokinetic (PK) sampling

DETAILED DESCRIPTION:
A randomized, parallel arm, double-masked, placebo-controlled Phase 3 study in at least 330 randomized subjects, evaluating the safety and efficacy of Nyxol in subjects with pharmacologically-induced mydriasis.

Following the successful completion of screening, each subject will be stratified by eye color and then simultaneously be randomized to mydriatic agent (unmasked) and treatment (masked). Treatment randomization will be 2:1, Nyxol or placebo (vehicle). Stratification by iris color will be 1:1, light or dark rides. The mydriatic agent randomization will be 3:1:1 (2.5% phenylephrine, 1% tropicamide, and Paremyd).

At the treatment visit, subjects who have been randomized and stratified by iris color (1:1 [light/dark]) will receive one of three approved mydriatic agents approximately 1 hour prior to receiving study treatment. Measurements will be measured before (-1 hour /baseline) and 60 minutes after (maximum/0 minutes) the mydriatic agent instillation in each eye (i.e. right before the study treatment is administered), and at 30 minutes, 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, and 6 hours after treatment dosing. Measurements will include pupil diameter (PD), distance and near visual acuity (VA), accommodation, and redness in each eye.

Blood sampling for Nyxol PK measurements will be conducted in a subset of approximately 30 adult subjects at approximately two select study sites.

At the Follow-Up Visit, which is 1 day after Visit 1, measurements will again be recorded 24 hours after treatment dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 12 years of age
2. Ability to comply with all protocol-mandated procedures independently and to attend all scheduled office visits

Exclusion Criteria:

1. Clinically significant ocular disease as deemed by the Investigator (eg, glaucoma, corneal edema, uveitis, severe keratoconjunctivitis sicca) that might interfere with the study
2. Unwilling or unable to discontinue use of contact lenses at screening until study completion
3. Unwilling or unable to suspend use of topical medication at screening until study completion
4. Ocular trauma, ocular surgery, or non-refractive laser treatment within the 6 months prior to screening
5. Use of any topical prescription or over-the-counter (OTC) ophthalmic medications of any kind within 7 days of screening, with the exception of lid scrubs with OTC products (eg, OCuSOFT® lid scrub, SteriLid®, baby shampoo, etc.)
6. Recent or current evidence of ocular infection or inflammation in either eye (such as current evidence of clinically significant blepharitis, conjunctivitis, or keratitis). Subjects must be symptom-free for at least 7 days prior to screening
7. Closed or very narrow-angle that in the Investigator's opinion is potentially occludable if the subject's pupil is dilated
8. Prior participation in a study involving the use of Nyxol for the reversal of mydriasis
9. Known hypersensitivity or contraindication to α- and/or β-adrenoceptor antagonists
10. Clinically significant systemic disease (eg, uncontrolled diabetes, myasthenia gravis, cancer, hepatic, renal, endocrine, or cardiovascular disorders) that might interfere with the study
11. Participation in any investigational study within 30 days prior to screening
12. Resting heart rate (HR) outside the normal range (50-110 beats per minute) at the Screening Visit.
13. Hypertension with resting diastolic blood pressure (BP)>105 mmHg or systolic BP > 160 mmHg at the Screening Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Clinical Site 10, Newport Beach, California
  - Clinical Site 12, Westminster, California
  - Clinical Site 9, Delray Beach, Florida
  - Clinical Site 8, Longwood, Florida
  - Clinical Site 6, Morrow, Georgia
  - Clinical Site 1, Roswell, Georgia
  - Clinical Site 13, Lake Villa, Illinois
  - Clinical Site 5, Pittsburg, Kansas
  - Clinical Site 2, Bloomington, Minnesota
  - Clinical Site 15, Garner, North Carolina
  - Clinical Site 4, Athens, Ohio
  - Clinical Site 14, Shrewsbury, Pennsylvania
  - Clinical Site 7, Warwick, Rhode Island
  - Clinical Site 11, Sioux Falls, South Dakota
  - Clinical Site 3, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phentolamine Ophthalmic Solution Vehicle: 2 drops in study eye and 1 drop in non-study eye, administered 1 hour post pharmacologically-induced mydriasis
  Phentolamine Ophthalmic Solution Vehicle: Phentolamine Ophthalmic Solution Vehicle
Period: Overall Study
Arm/Group | Phentolamine Ophthalmic Solution Vehicle | Phentolamine Ophthalmic Solution 0.75%
Started | 124 | 244
Completed | 124 | 244
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 244 | 124 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (15.61) | 35.6 (17.58) | 34.6 (16.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 65 | 217
  Male | 92 | 59 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 9 | 30
  Not Hispanic or Latino | 223 | 115 | 338
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 22 | 9 | 31
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 38 | 21 | 59
  White | 179 | 93 | 272
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 244 | 124 | 368

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects' Study Eyes With Pupil Diameter Returning to Baseline
Description: Percentage of subjects' study eyes returning to less than or equal to 0.2 mm from baseline pupil diameter
Time Frame: 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 244 | 124
Participants
  Returning to <= 0.2mm of Baseline | 142 | 7
  Not returning to <= 0.2mm of Baseline | 102 | 117

2. Secondary Outcome: Percent of Subjects' Study Eyes With Pupil Diameter Returning to Baseline
Description: Percentage of subjects' study eyes returning to less than or equal to 0.2 mm from baseline pupil diameter
Time Frame: 30 minutes to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 244 | 124
Participants
  30 minutes: Returning to <=0.2 mm of Baseline | 10 | 5
  30 minutes: Not returning to <=0.2 mm of Baseline | 234 | 119
  60 minutes: Returning to <=0.2 mm of Baseline | 103 | 3
  60 minutes: Not returning to <=0.2 mm of Baseline | 141 | 121
  90 minutes: Returning to <=0.2 mm of Baseline | 142 | 7
  90 minutes: Not returning to <=0.2 mm of Baseline | 102 | 117
  2 Hours: Returning to <=0.2 mm of Baseline | 162 | 9
  2 Hours: Not returning to <=0.2 mm of Baseline | 82 | 115
  3 Hours: Returning to <=0.2 mm of Baseline | 193 | 17
  3 Hours: Not returning to <=0.2 mm of Baseline | 51 | 107
  4 Hours: Returning to <=0.2 mm of Baseline | 210 | 21
  4 Hours: Not returning to <=0.2 mm of Baseline | 34 | 103
  6 Hours: Returning to <=0.2 mm of Baseline | 221 | 44
  6 Hours: Not returning to <=0.2 mm of Baseline | 23 | 80
  24 Hours: Returning to <=0.2 mm of Baseline | 218 | 89
  24 Hours: Not returning to <=0.2 mm of Baseline | 26 | 35

3. Secondary Outcome: Pupil Diameter (Change From Max)
Description: Change (mm) from maximum pharmacologically-induced mydriatic pupil diameter (0 minutes)
Time Frame: 30 minutes to 24 hours
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 244 | 124
millimeters
  30 Minutes | -0.109 (0.7104) | 0.092 (0.5335)
  60 Minutes | -1.457 (1.0825) | -0.059 (0.5775)
  90 Minutes | -2.157 (1.1911) | -0.284 (0.5852)
  2 Hours | -2.478 (1.1453) | -0.488 (0.6807)
  3 Hours | -2.917 (1.1721) | -0.987 (0.7932)
  4 Hours | -3.078 (1.1578) | -1.261 (0.8615)
  6 Hours | -3.267 (1.2743) | -1.755 (1.0205)
  24 Hours | -3.134 (1.3607) | -2.313 (1.3607)

4. Secondary Outcome: Percent of Subjects With Unchanged Accommodation From Baseline
Description: Percentage of subjects with unchanged accommodation from baseline (-1 hour)
Time Frame: 90 minutes to 6 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 244 | 124
Participants
  90 Minutes: Unchanged from Baseline | 155 | 65
  90 Minutes: Changed from Baseline | 89 | 59
  2 Hours: Unchanged from Baseline | 165 | 66
  2 Hours: Changed from Baseline | 79 | 58
  3 Hours: Unchanged from Baseline | 186 | 81
  3 Hours: Changed from Baseline | 58 | 43
  6 Hours: Unchanged from Baseline | 204 | 86
  6 Hours: Changed from Baseline | 40 | 38

5. Secondary Outcome: Change From Baseline in Best-Corrected Distance Visual Acuity (BCDVA) Under Normal Photopic Lighting Without Glare Conditions
Description: Change from Baseline in best-corrected distance visual acuity (BCDVA) under normal photopic lighting without glare conditions
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
Number analyzed (Participants) | 244 | 124
letters | 0.3 (3.73) | -0.2 (4.64)

ADVERSE EVENTS:
Time Frame: 2 Days
Arm/Group | Phentolamine Ophthalmic Solution 0.75% | Phentolamine Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/124
Other Adverse Events (participants affected / at risk) | 43/244 | 0/124
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phentolamine Ophthalmic Solution 0.75% (N=244) | Phentolamine Ophthalmic Solution Vehicle (N=124)
Conjunctival Hyperaemia (Eye disorders) | 26 | 0
Instillation site erythema (General disorders) | 9 | 0
Dysgeusia (Nervous system disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT05134974/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT05134974/SAP_002.pdf